CLINICAL TRIAL: NCT04900623
Title: Risk-adapted Therapy in HPV+ Oropharyngeal Cancer Using Circulating Tumor (ct)HPV DNA Profile - The ReACT Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonathan Schoenfeld, MD, MPH (Other)
Collaborators: Naveris (Unknown)
Responsible Party: Sponsor-Investigator, Jonathan Schoenfeld, MD, MPH, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-191
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HPV-Associated Oropharyngeal Squamous Cell Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma; HPV-Mediated (P16-Positive) Oropharyngeal Carcinoma by AJCC V8 Stage; HPV-Related Squamous Cell Carcinoma; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; HPV-Mediated (P16-Positive) Oropharyngeal Carcinoma by AJCC V8 Clinical Stage; HPV-Mediated (P16-Positive) Oropharyngeal Carcinoma by AJCC V8 Pathologic Stage
Keywords: HPV-Associated Oropharyngeal Squamous Cell Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma; HPV-Mediated (P16-Positive) Oropharyngeal Carcinoma by AJCC V8 Pathologic Stage; HPV-Mediated (P16-Positive) Oropharyngeal Carcinoma by AJCC V8 Clinical Stage; Pathologic Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiotherapy; Radiotherapy, Intensity-Modulated; Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- LOW RISK RT (ALONE OR WITH SOC CHEMO (Experimental): The research study procedures include: screening for eligibility, and study treatments including evaluations and follow-up visits
  * NavDx HPV ctDNA Testing: Blood will be collected and shared with an outside lab for analysis (less than 10 mL of blood or about 2 teaspoons). The results of this test will determine what radiation dose received . The specimens will be de-identified. The specimens will be banked for future use.
  * Radiation Therapy: Lower risk participants will receive a lower dose and treatment will only last 5-6 weeks.
  * Chemotherapy: Chemotherapy and radiation therapy are both considered standard treatments for your type of cancer. The study doctor will decide whether or not chemotherapy with radiation and the type of chemotherapy.
    * Bolus Cisplatin: Infused every 21 days for up to 2 or 3 doses.
    * Weekly Cisplatin or Carboplatin with Paclitaxel: Infused weekly during radiation therapy
  Interventions: Device: NavDx HPV ctDNA Testing; Radiation: Radiotherapy; Drug: Chemotherapy drug
- INTERMEDIATE RISK RT (ALONE OR WITH SOC CHEMO (Experimental): The research study procedures include: screening for eligibility, and study treatments including evaluations and follow-up visits
  * NavDx HPV ctDNA Testing: Blood will be collected and shared with an outside lab for analysis (less than 10 mL of blood or about 2 teaspoons). The results of this test will determine what dose of radiation received. The specimens will be de-identified. The specimens will be banked for future use.
  * Radiation Therapy: Higher risk participants will receive standard radiation dose for up to 7-8 weeks
  * Chemotherapy: Chemotherapy and radiation therapy are both considered standard treatments for your type of cancer. The study doctor will decide whether or not chemotherapy with radiation and the type of chemotherapy.
    * Bolus Cisplatin: Infused every 21 days for up to 2 or 3 doses.
    * Weekly Cisplatin or Carboplatin with Paclitaxel: Infused weekly during radiation therapy
  Interventions: Device: NavDx HPV ctDNA Testing; Radiation: Radiotherapy; Drug: Chemotherapy drug

INTERVENTIONS:
Device: NavDx HPV ctDNA Testing — Blood will be collected and shared with an outside lab for analysis. This test will be done at Week 4 and at End of Treatment. This test will be done at at End of Treatment and in follow-up at 3, 6, 9, and 12 months after completing the study treatment. In years 2 and 3 after treatment, the test will be collected every 6 months or twice a year. The specimens will be identifiable. The specimens will be banked for future use.
  Other Names: NavDx
Radiation: Radiotherapy — Radiation Therapy (administered daily, Monday-Friday). Higher risk participants will receive standard radiation dose for up to 7-8 weeks. Lower risk participants will receive a lower dose and treatment will only last 5-6 weeks.
  Other Names: Intensity-modulated radiotherapy (IMRT); Proton beam radiotherapy
Drug: Chemotherapy drug — Chemotherapy and radiation therapy are both considered standard treatments
  * Bolus Cisplatin: Infused every 21 days for up to 2 or 3 doses.
  * Weekly Cisplatin or Carboplatin with Paclitaxel: Infused weekly during radiation therapy.
  Other Names: Bolus Cisplatin; Cisplatin; Carboplatin with Paclitaxel

SUMMARY:
This research is being conducted to understand if treatment can be tailored for participants with HPV-related oropharynx cancers using both clinical features (stage of the tumor, smoking status) combined with an investigational HPV blood test.

The names of the test and treatments involved in this study are:

* NavDx® HPV ctDNA testing (HPV blood test)
* Radiation therapy
* Chemotherapy: Cisplatin, or Carboplatin and Paclitaxel (not all participants receive any or all of these agents)

DETAILED DESCRIPTION:
This research study involves HPV DNA testing (a blood test that measures the levels of DNA from the human papillomavirus in the bloodstream which investigator think sheds from the cancer itself), radiation therapy, and chemotherapy for some participants.

The research study procedures includes: screening for eligibility, and study treatments including evaluations and follow-up visits.

The names of the test and treatments involved in this study are:

* NavDx® HPV ctDNA testing (HPV blood test)
* Radiation therapy: Radiation therapy alone or combined with chemotherapy is considered a standard treatment for this disease. The investigators are researching the effectiveness of reducing the radiation doses and, in some cases, also reducing the chemotherapy dose for certain participants with favorable clinical characteristics and with certain HPV blood test results.
* Chemotherapy: Cisplatin, or Carboplatin and Paclitaxel (not all participants receive any or all of these agents)
* Study treatment will for up to 7 weeks and participants will be followed for 5 years from the beginning of the study.
* It is expected that about 145 people will take part in this research study.

The HPV ctDNA levels will be measured using a blood test called NavDx®, which will be provided free of charge from the company NAVERIS. ctDNA testing refers to circulating tumor (ct)DNA or measuring DNA fragments floating in the bloodstream that are released from the cancer cells. This testing has shown promise in early detection of cancer recurrence in several solid tumor types (including colorectal, urothelial, and breast cancer). Additionally, recent studies have shown a connection between baseline ctDNA levels and disease risk.

The U.S. Food and Drug Administration (FDA) has not approved NavDx® as a method for guiding treatment decision-making, but this is an important part of this research study. While the NavDx® assay is investigational, it is performed in a Clinical Laboratory Improvement Amendment (CLIA) certified clinical laboratory and is currently available as a clinical tool for measuring HPV ctDNA levels in some cancer patients. CLIA regulations include federal standards applicable to all United States facilities or sites that test human specimens for health assessment or to diagnose, prevent, or treat disease

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. Radiation therapy alone or combined with chemotherapy is considered a standard treatment for this disease. The investigators are researching the effectiveness of reducing the radiation doses and, in some cases, also reducing the chemotherapy dose for certain participants with favorable clinical characteristics and with certain HPV blood test results.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following eligibility criteria at the time of screening to be eligible to participate in the study:
* Subject must have histologically or cytologically confirmed, stage I, II, or III (N3 disease excluded), HPV associated oropharyngeal (tongue base or tonsil) squamous cell carcinoma, as defined by 2017 American Joint Committee on Cancer (AJCC), 8th edition staging.

  -- Patients with HPV-associated disease of unknown primary (cT0) are eligible
* HPV status should be confirmed on tissue biopsy or cytologic sample by any of the following:

  * Immunohistochemical staining for p16 with ≥70% expression
  * Confirmatory DNA testing (PCR or ISH) for high-risk subtype
* Willing to provide blood and tissue from a diagnostic biopsy and blood samples before, during, and after treatment.
* Detectable HPV ctDNA blood sample at baseline, prior to treatment, using the NavDx® assay that detects HPV subtype 16
* Age 22 years or older
* ECOG performance status ≤ 2
* Participants should have adequate organ and marrow function if they are to receive chemotherapy (cisplatin, or carboplatin and paclitaxel) with radiation concurrently as determined by standard institutional guidelines and investigator preference (parameters suggested below).

  * absolute neutrophil count (ANC) ≥ 1000
  * platelet count ≥ 100,000
  * total bilirubin of 1.5 or less
  * creatinine of 1.6 or less (or a CrCl ≥50 mL/min) per institutional standards.
* Planning to receive non-surgical management for HPV+ oropharyngeal cancer
* Ability to understand and the willingness to sign a written informed consent document.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of (chemo)radiation therapy. "Women of childbearing potential (WOCBP)" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level above 40 mIU/mL.
* Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 1 month after treatment. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception.

Exclusion Criteria:

* Patients with AJCC 2017 8th edition stage IVC (metastatic) disease; or patients with fixed cervical nodal disease suggesting extranodal extension or N3 disease as suggested by lymph nodes measuring >6 cm.
* Subject who has had prior radiation and/or chemotherapy for head and neck cancer.
* Any history of oncologic surgical resection (transoral robotic surgery, TORS) or oncologic neck dissection prior to undergoing definitive RT or chemoradiation. Note: prior tonsillectomy as part of identification of the primary tumor site or biopsy and excisional nodal biopsy is/are acceptable provided the patient would be standardly treated to definitive treatment doses of therapy off protocol. Patients with HPV-associated unknown primary should not have undergone a neck dissection to be eligible.
* Undetectable baseline HPV ctDNA result by NavDx® testing or detectable baseline HPV ctDNA result for subtypes 18, 31, 33, or 35.
* Pregnant or lactating women.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, and low risk prostate adenocarcinoma being managed with active surveillance. A history of another separate malignancy in remission without evidence of active disease is permitted if chance3 of recurrence is thought to be low.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival 2 Years | 2 Years
  Progression-free survival (PFS) is defined as the time from the date of study registration to first invasive local, regional, distant progression, or death due to any cause. Participants alive without progression are censored at date of last disease evaluation

SECONDARY OUTCOMES:
Overall Survival at 2 Years | 2 Years
  Defined as the time from study registration to death due to any cause, or censored at date last known alive.
Rate of Distant Failure | every 12 weeks (or 3 months) from the time of therapy completion for years 1 and 2, and every 24 weeks (or 6 months) from the time of therapy completion in year 3.
  Distant metastatic-free survival (DMFS) is defined as the time from confirmed disease response (CR/PR) to the earlier of the first occurrence of distant or metastatic disease, or death due to any cause. Participants alive without distant or metastatic progression are censored at date of last disease evaluation.
Best Overall Response | every 12 weeks (or 3 months) from the time of therapy completion for years 1 and 2, and every 24 weeks (or 6 months) from the time of therapy completion in year 3.
  The best response recorded from the start of the treatment until disease progression or recurrence, with documentation of local (primary site) or regional (neck lymph node) disease clearance being of interest. Clinical or radiographic evidence of progressive locoregional disease beyond 12 weeks (or 3 months) from the end of treatment should be documented and ideally confirmed by locoregional or distant disease biopsy, neck dissection, or salvage surgery. CT or MRI (of head and neck region, with chest CT), or PET-CT may be used as radiographic evaluation of overall disease status.
Score Change FACT-H&N survey data | baseline up to 5 years
  The self-administered Functional Assessment of Cancer Therapy - Head & Neck Cancer (FACT-HN) questionnaire consists of FACT-G, a cancer specific QOL questionnaire that includes 27 questions in 4 domains - physical, social, emotional, and function, and a 12-time H&N cancer-specific modules. Each item is rated on a 0 to 4 scale. Higher scores represent better Quality of Life. A clinically significant change in score on this instrument is represented by an increase of 6 units or decrease of 12 units
Safety and Toxicity | 6 and 12 months after protocol therapy
  Evaluated by measuring feeding tube rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Schoenfeld, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu